CLINICAL TRIAL: NCT05662007
Title: Scapular Kinematics of Asymptomatic Young Swimmers During Dynamic Shoulder Elevation
Brief Title: Scapular Kinematics of Young Swimmers
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ferhat Öztürk, Principal Investigator, Hacettepe University
Other Study IDs: GO20/240
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Scapula Injuries
Keywords: swimmers; scapula; kinematic; motion asymmetries; three dimensional

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young swimmers group
- Healthy Control Group

INTERVENTIONS:
Other:  — no intervention

SUMMARY:
The aim of this study was to (a) compare the scapular kinematics of asymptomatic swimmers and healthy non-athletes and to (b) compare the scapular kinematics of the dominant and non-dominant shoulders in asymptomatic young swimmers.

DETAILED DESCRIPTION:
This cross-sectional study included 27 volunteered asymptomatic young swimmers (mean age: 12.7 yrs) with at least 3 years of experience in a professional swimming club and 22 healthy non-athletes (mean age: 11.5 yrs). 3D scapular kinematics were evaluated at 0°, 30º, 60º, 90º, and 120º with the electromagnetic tracking system during bilateral arm elevation and lowering on the scapular plane. The differences in the scapular kinematics of the dominant and the non-dominant side in both groups were analyzed with 2 by 8 Mixed Model ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* Absence of shoulder pain in the last 6 months,
* No discomfort in the shoulder joint during swimming,
* Use of symmetrical breathing patterns in training competitions

Exclusion Criteria:

* Participants with a history of upper extremity injury (dislocation, fracture, muscle strain, etc.),
* Pain in clinical tests (Hawkins and Neer),
* Those who did not attend training regularly.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This cross-sectional study included volunteer young swimmers with at least 3 years of experience in a professional swimming club and healthy non-athletes participants. The swimmer training program includes swimming training 6 days a week (10 hours in total), and 3 land training (3 hours in total) including a general strengthening program (strength of the posterior shoulder musculature, core, squats, pull-ups, etc.) and stretching the anterior shoulder musculature.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Scapular Kinematic | one year
  3D scapular kinematics were evaluated at 0°, 30º, 60º, 90º, and 120º with the electromagnetic tracking system during bilateral arm elevation and lowering on the scapular plane. The differences in the scapular kinematics of the dominant and the non-dominant side in both groups were analyzed with 2 by 8 Mixed Model ANOVA.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No